CLINICAL TRIAL: NCT04747431
Title: A Phase 1b Open-Label, Multicenter, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacodynamic Effects of a Single Dose of PBFT02 Delivered Into the ICM of Adults With FTD and Mutations in the GRN or C9ORF72 Genes
Brief Title: A Study of PBFT02 in Participants With FTD and Mutations in the Granulin Precursor (GRN) or C9ORF72 Genes
Acronym: upliFT-D
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Passage Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBFT02-001; 2020-004499-17 (EudraCT Number)
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Frontotemporal Dementia; FTD; FTD-GRN; Dementia Frontotemporal; C9orf72
Keywords: frontotemporal dementia; Progranulin Mutations; FTD-GRN; Gene Therapy; Dementia Gene Therapy; AAV1; Fronto-temporal Dementia; C9orf72
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain; Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: Open-label, multi-center, dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Drug: PBFT02 Dose 1; Single dose of PBFT02, via intra cisterna magna
  *GC/g: gene copy per gram of estimated brain weight
  Interventions: Drug: PBFT02
- Cohort 2, 3, 4 and 5 (Experimental): Drug: PBFT02 Dose 1 or 2; Single dose of PBFT02, via intra cisterna magna
  *GC/g: gene copy per gram of estimated brain weight
  Interventions: Drug: PBFT02

INTERVENTIONS:
Drug: PBFT02 — PBFT02

SUMMARY:
PBFT02 is a gene therapy for frontotemporal dementia intended to deliver a functional copy of the GRN gene to the brain. This study will assess the safety, tolerability and efficacy of this treatment in patients with frontotemporal dementia and mutations in the granulin precursor (GRN) or chromosome 9 open reading frame 72 (C9ORF72) genes

DETAILED DESCRIPTION:
PBFT02 is an adeno-associated viral vector serotype 1 carrying GRN, the gene encoding for human progranulin, formulated as a solution for injection into the cisterna magna. This is a global interventional, multicenter, open-label, single-arm study of PBFT02 delivered as a one-time dose administered into the cisterna magna to participants with FTD-GRN or C9orf72. Participants aged ≥ 35 and ≤ 75 years with early symptomatic FTD-GRN or with symptomatic FTD-C9orf72 may be enrolled into the study.

PBFT02 will be studied in three cohorts of FTD-GRN participants and two cohorts of FTD-C9orf72 participants.

This is a 5-year study, with a 2-year main study, followed by a 3-year safety extension.

ELIGIBILITY:
Inclusion Criteria:

1. Documented to be a pathogenic carrier of GRN or C9orf72 mutation
2. Clinical diagnosis of frontotemporal dementia
3. Have a reliable informant / caregiver (and back-up informant / caregiver) who personally speaks with or sees the subject at least weekly
4. Living in the community (i.e., not in a nursing home); assisted living may be permitted at the discretion of the investigator

Exclusion Criteria:

1. Classification of the GRN mutation as "not pathogenic," "likely benign variant," "benign variant," or "pathogenic nature unclear" (FTD- GRN Cohorts 1-3) or C9orf72 HRE length ≤ 30 (FTD-C9orf72 Cohorts 4-5).
2. Previous treatment with any gene therapy. Any other therapies with the potential to alter PGRN levels must be washed out for at least 5 half-lives prior to entry into this study
3. Homozygous GRN mutation carrier (FTD-GRN Cohorts 1-3) or homozygous C9orf72 mutation carrier (FTD-C9orf72 Cohorts 4-5).
4. Rosen-modified Hachinski Ischemic Scale score > 7
5. Known presence of a structural brain lesion (eg, tumor, cortical infarct) that could reasonably explain symptoms in a symptomatic subject
6. Known presence of an AD-causing mutation in PSEN1, PSEN2 or APP based on genetic testing history (if performed)
7. Previous history of Korsakoff encephalopathy, severe alcohol or substance dependence (within 5 years of onset of dementia), except where onset of increased alcohol consumption occurs at the time of FTD disease onset
8. History of untreated vitamin B12 deficiency
9. Presence of untreated hypothyroidism (thyroid stimulating hormone [TSH] > ULN and free T4 < LLN)
10. eGFR ≤ 30 ml/min (as calculated using the CKD-EPI equation)
11. Alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 2 × ULN, or total bilirubin > ULN)
12. Respiratory failure that requires supplemental oxygen, tracheostomy, or reliance on non-invasive ventilation for >2 hours during waking hours
13. Inability to provide full consent or the lack of a legally authorized caregiver with adequate contact who can provide consent
14. Any contraindication to MRI or lumbar puncture (LP) (eg, local infection, history of thrombocytopenia, coagulopathy)
15. Any contraindication to the ICM administration procedure
16. Medical conditions or laboratory or vital sign abnormalities that would increase risk of complications from ICM injection, anesthesia, LP, and/or MRI (e.g., fever, hypoxia, tachycardia, or evidence of active infection)
17. Immunocompromised status
18. Peripheral axonal sensory neuropathy
19. Receipt of a vaccine within 14 days of dosing
20. A positive test result for human immunodeficiency virus (HIV), human T cell leukemia virus (HTLV) type 1 or type 2, or Hepatitis B or C; a Mycobacterium tuberculosis positive test within 1 year of or determined at screening
21. Malignant neoplasia (except localized skin cancer) or a documented history of hereditary cancer syndrome
22. Any concurrent disease that, in the opinion of the investigator, may cause cognitive impairment unrelated to GRN or C9orf72 mutations, including other causes of dementia, neurosyphilis, hydrocephalus, stroke, small vessel ischemic disease, uncontrolled hypothyroidism, or vitamin deficiency
23. Current or recent history of clinically significant suicidal ideation within the past 6 months
24. For women of childbearing potential, a positive serum pregnancy test at the screening visit, a positive serum result on Day 1 prior to administration of the investigational product, or unwillingness to have additional pregnancy tests during the study. Women of childbearing potential must use a highly effective method of birth control or engage in abstinence until 90 days postdose
25. Women who are breastfeeding
26. For sexually active men, unwillingness to use a medically accepted method of double-barrier contraception (such as a condom/diaphragm used with spermicide) or engage in abstinence from the date of screening until 90 days postdose
27. Any condition (eg, history of any disease, evidence of any current disease, any finding upon physical examination, or any laboratory abnormality) that, in the opinion of the investigator, would put the subject at undue risk or would interfere with evaluation of the investigational product or interpretation of subject safety or study results
28. Any acute illness requiring hospitalization within 30 days of enrollment
29. Failure to meet the protocol-specified coagulation test criteria:

    * Platelet count > 100,000 per uL
    * INR < 1.5
    * aPTT < 40 seconds
30. Use of anticoagulants in the 2 weeks prior to screening
31. Hypersensitivity or contraindications to corticosteroid use
32. Known or suspected intolerance or hypersensitivity to PBFT02 or any of its ingredients or to closely related compounds
33. Any condition expected to increase risk of thrombosis
34. Hypersensitivity or contraindications to apixaban

    Additional Criteria for FTD-C9orf72 (Cohorts 4-5) ONLY: Presence of concurrent ALS is permitted provided the following criteria are NOT met:
35. ALSFRS-R < 35 at screening.
36. SVC < 75% of predicted normal adjusted for sex, age, and height (from the sitting position).
37. Bulbar-onset ALS.
38. Current or anticipated need, in the opinion of the Investigator for a diaphragm pacing system (DPS) during the study period.
39. If taking riluzole or edaravone, participant's dose has not been stable for ≥ 30 days prior to Day 1 and/or dose adjustments are anticipated before the Day 60 study visit.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related AEs and SAEs | Up to 5 years (multiple visits)
  Assess the number of treatment-related adverse events (AEs) and serious adverse events (SAEs)
Change in Nerve Conduction Velocity and Amplitude from Baseline on Nerve Conduction Studies | From baseline to 5 years (multiple visits)
  Assess changes in nerve conduction velocity in the distal segments of the sural, radial, and median sensory nerves and peroneal motor nerve as measured on conventional nerve conduction studies.
Change in Cellular and Humoral Response Against the Vector and Transgene in Serum | From baseline to 5 years (multiple visits)
  Assess ELISpot and antibody titers against AAV1 and against human progranulin

SECONDARY OUTCOMES:
Change from baseline in CSF and plasma PGRN levels | From baseline to 5 years (multiple visits)
  Assess effect of treatment with PBFT02 on CSF and plasma PGRN levels following administration of a single ICM dose.
Change from baseline in plasma and CSF neurofilament light chain (NfL) levels | From baseline to 5 years (multiple visits)
  Assess the effect of treatment with PBFT02 on PGRN level in CSF and plasma
Change in Brain anatomy as assessed by MRI | From baseline to 5 years (multiple visits)
  Assess the effect of treatment with PBFT02 on Brain volume, white matter integrity, and cortical thickness as assessed by MRI
Change in FTLD disease progression | From baseline to 5 years (multiple visits)
  Assess changes in the Clinical Dementia Rating Scale for Frontotemporal Lobar Degeneration plus National Alzheimer's Coordinating Center FTLD Behavior & Language Domains (CDR® plus NACC FTLD SB)
Change in ALS disease progression in participants with FTD C9orf72 | From baseline to 5 years (multiple visits)
  Assess changes in ALS disease progression using the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R), percent predicted slow vital capacity (SVC) and in muscle strength as measured by handheld dynamometry (HHD)
Change in vital status | From Baseline to 5 years (multiple years)
  Assess the impact of PBFT02 on survival

CONTACTS AND LOCATIONS:
Overall Officials: Tiffini Voss, MD, PhD, Study Director — Passage Bio, Inc.
Locations (10):
- United States (4):
  - Michigan Alzheimer's Disease Center, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas at Houston, Houston, Texas
- Eastern Health-Box Hill Hospital, Melbourne, Victoria, Australia
- Brazil (2):
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (UFMG), Minas Gerais
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo (HCFMUSP), São Paulo
- Canada (2):
  - University of Toronto, Toronto Western Hospital, Toronto, Ontario
  - Montreal Neurological Institute-Hospital, Montreal, Quebec
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No